CLINICAL TRIAL: NCT00000217
Title: Pharmacotherapy and Intensive Treatment of Drug Abuse
Brief Title: Pharmacotherapy and Intensive Treatment of Drug Abuse - 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Kansas (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: University of Kansas Medical Center (Other)
Purpose: Treatment
Other Study IDs: NIDA-06954-1; R18DA006954 (NIH); R18-06954-1
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-04

CONDITIONS: Cocaine-Related Disorders; Substance-Related Disorders
Keywords: drug abuse
MeSH Terms: conditions — Cocaine-Related Disorders; Substance-Related Disorders | interventions — Carbamazepine

INTERVENTIONS:
Drug: Carbamazepine

SUMMARY:
The purpose of this study is to evaluate desipramine and carbamazepine in reducing cocaine craving; increase outpatient treatment capacity and evaluate their incidence of psychiatric disorders.

ELIGIBILITY:
Please contact site for information.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 1990-09; Primary Completion 1996-10 (Actual)

PRIMARY OUTCOMES:
Drug use
Effectiveness of medication
Level of pharm
Retention
Depression, anxiety

CONTACTS AND LOCATIONS:
Overall Officials: William Haning, M.D., Principal Investigator — University of Kansas
Locations (1):
- University of Kansas, Kansas City, Missouri, United States

REFERENCES:
- [Background] J Addictive Dis. 13; 1994